CLINICAL TRIAL: NCT03108040
Title: Evaluation of Non Invasive Fetal Cardiac Functions and Fetal Arterial&Venous Doppler Study in Intrauterine Growth Restriction as Predictive Parameters of Perinatal Outcome
Brief Title: Evaluation of Fetal Cardiac Function and Vascular Hemodynamics in Intrauterine Growth Restriction
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sief el eslam Ahmed Ali, Principal investigator, Assiut University
Other Study IDs: AUN80
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Fetal Hypoxia
MeSH Terms: conditions — Fetal Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Intrauterine growth restriction (IUGR) is one of the major contributors to perinatal mortality and morbidity and is characterized by complex hemodynamic changes involving placental and fetal arterial, cardiac and venous circulations .However, the temporal sequence of these modifications in relation to other hemodynamic changes of the fetal arterial and venous circulations is unknown.

The aim of this study was to evaluate cardiac function and other hemodynamic changes in a group of fetuses with IUGR and clinical impact on perinatal outcome .

ELIGIBILITY:
Inclusion Criteria:

* Singleton fetus with normal fetal anatomy documented a detailed sonogram.
* Fetal abdominal circumference <5th percentile for gestational age.
* Evidence of placental insufficiency documented by an elevated umbilical artery pulsatility index (UA-PI) by reference ranges.

Exclusion Criteria:

* evidence of fetal infection
* chorioamnionitis
* fetal anomalies
* abnormal fetal karyotype
* patient withdrawal from the study and/or unavailability for follow-up.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: observational study conducted at academic perinatalcenter that investigates relationships between antenatal testing parameters and outcome in IUGR fetuses Patients who give written consent to participate in the study undergo a uniform antenatal assessment protocol that includes umbilical artery (UA), middle cerebral artery (MCA) and ductus venosus (DV) Doppler ultrasound studies as well as detailed fetal echocardiography and five-component biophysical profile score.
  - Criteria for study eligibility are:
  * Singleton fetus with normal fetal anatomy documentedon a detailed sonogram.
  * Fetal abdominal circumference <5th percentile forgestational age.•
  * Evidence of placental insufficiency documented by an elevated umbilical artery pulsatility index (UA-PI) by reference ranges.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Myocardial performance index | 5 minutes
  Ratio between isovolumetric time to ejection time
Aortic isthmus flow index | 5 minutes
  Aortic isthmus flow index = Ratio of (systolic velocity time integral+diastolic velocity time integral) / systolic velocity time integral
Cerebroplacental ratio | 5 minutes
  cerebroplacental ratio = Rtio middle cerebral artery pulsatility index / umbilical artery pulsatility index
Preload Index in inferior vena cava | 5 minutes
  Preload Index in inferior vena cava = ratio of peak systolic velocity in atrial contraction /peak systolic velocity ventricular systole

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Fetal Cair Unit - Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided